CLINICAL TRIAL: NCT03509948
Title: A Phase 1 Open Label, Randomized, Two-Way Crossover Study in Healthy Smokers to Investigate the Effect of Food on the Bioavailability of Cytisine in a New Formulation
Brief Title: A Study in Healthy Smokers to Investigate the Effect of Food on the Bioavailability of Cytisine in a New Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CYT-07
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Schedule A: Fed Then Fasted (Experimental): Schedule A (6 participants):
  * Period 1: cytisine (2 x 1.5 mg tablets) will be administered 30 minutes after the start of a high fat breakfast (fed state)
  * Period 2: cytisine (2 x 1.5 mg tablets) will be administered after an overnight fast of at least 10 hours (fasting state)
  Interventions: Drug: cytisine
- Schedule B: Fasted Then Fed (Experimental): Schedule B (6 participants):
  * Period 1: cytisine (2 x 1.5 mg tablets) will be administered after an overnight fast of at least 10 hours (fasting state)
  * Period 2: cytisine (2 x 1.5 mg tablets) will be administered 30 minutes after the start of a high fat breakfast (fed state)
  Interventions: Drug: cytisine

INTERVENTIONS:
Drug: cytisine — cytisine 1.5 mg film-coated tablets
  Other Names: Tabex

SUMMARY:
This will be an open-label, randomised, 2-treatment period, single-dose crossover study to determine the comparative bioavailability and renal elimination following single-dose administration of 3.0 mg cytisine in healthy smokers under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

To be Confirmed at Screening

1. Subject is current cigarette smoker.
2. Healthy males and females between 18 and 55 years of age.

   1. If a female subject of child bearing potential, a negative pregnancy test at screening and admission and willing to use an effective method of contraception (unless of non-childbearing potential or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of cytisine.
   2. If a female subject of non-child bearing potential, a negative pregnancy test at screening and admission. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status will be confirmed by demonstrating at screening that levels of follicle stimulating hormone (FSH) fall within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at Investigator's discretion following consultation with the Sponsor.
   3. If a male subject, willing to use an effective method of contraception (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of cytisine.
3. Subject with a body mass index (BMI) of 23-28 kg/m^2. BMI = body weight in kg / [height in m^2].
4. Subject with no clinically significant abnormal serum biochemistry or haematology values within 28 days before the first dose of cytisine.
5. Subject with negative urinary drugs of abuse screen, determined within 28 days before the first dose of cytisine (a positive result may be repeated at Investigator's discretion).
6. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
7. Subject with no clinically significant abnormalities in 12-lead ECG determined after minimum of 5 minutes in supine position within 28 days before the first dose of cytisine.
8. Subject with no clinically significant abnormalities in vital signs (systolic blood pressure between 90-140 mmHg, diastolic blood pressure (DBP) between 50 and 90 mmHg, and pulse rate (PR) between 40-100 bpm, measured on the dominant arm after minimum of 5 minutes in supine position) determined within 28 days before first dose of cytisine.
9. Subject must be available to complete the study (including post study follow-up) and comply with study restrictions.
10. Subject must provide written informed consent to participate in the study.

To be Re-Confirmed Prior to Dosing

1. Subject continues to meet all screening inclusion criteria (before the cytisine dose).
2. Subject has a negative urinary drugs of abuse screen (including alcohol).
3. Female subject has a negative urine pregnancy test.

Exclusion Criteria:

To be Confirmed at Screening

1. Known hypersensitivity/allergy reaction to varenicline, other cytisine-derivatives or any of the excipients in the Tabex formulation (cellulose, talc, magnesium).
2. History of severe hypersensitivity reactions to any other drugs.
3. History of any medical condition (e.g. gastrointestinal, renal or hepatic) or surgical condition (e.g. cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion).
4. Female subjects who are breast feeding.
5. Difficulty in donating blood on either arm or known history.
6. History of alcoholism or drug abuse within last 2 years.
7. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days (or 5 half-lives, whichever is longer) prior to the cytisine dose, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
8. Participated in any investigational drug clinical trial within the previous 3 months or a marketed drug trial within the previous 30 days prior to randomization on Day 1 of Period 1.
9. Donation of 450 mL or more blood or had history of significant blood loss due to any reason or had plasmapheresis within 3 months before the cytisine dose.
10. Any inability or difficulty in fasting.
11. Inability to communicate well with Investigators (i.e., language problem, poor mental development or impaired cerebral function).
12. Any other condition that the Principal Investigator considers making the subject unsuitable for this study.

To be Re-Confirmed Prior to Dosing:

1. Development of any exclusion criteria since screening.
2. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements since screening, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
3. Participation in a clinical study since the screening visit.
4. Donation of 450 mL or more blood since the screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezanul Abd Wahab, MD, Principal Investigator — Simbec Research Ltd (Simbec)
Locations (1):
- Simbec Research Ltd, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 mg Cytisine, Schedule A: Fed Then Fasted: * Period 1: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
- 3 mg Cytisine, Schedule B: Fasted Then Fed: * Period 1: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
Period: Overall Study
Arm/Group | 3 mg Cytisine, Schedule A: Fed Then Fasted | 3 mg Cytisine, Schedule B: Fasted Then Fed
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 3 mg Cytisine, Schedule A: Fed Then Fasted
  * Period 1: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
    3 mg Cytisine, Schedule B: Fasted Then Fed
  * Period 1: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state).
  * Period 2: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state).
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax)
Time Frame: Pre-dose (within 60 minutes prior to dosing), up to 48 hours post-dose on Days 1-5
Population: Pharmacokinetic (PK) Set: All randomized participants who received both doses of cytisine and had sufficient, protocol-compliant plasma concentration-time profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 3 mg Cytisine: Fed: Cytisine (2 x 1.5 mg tablets) administered 30 minutes after the start of a high fat breakfast (fed state)
- 3 mg Cytisine: Fasted: Cytisine (2 x 1.5 mg tablets) administered after an overnight fast of at least 10 hours (fasting state)
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
ng/mL | 26.2 (37.2) | 32.9 (23.7)
Statistical Analysis 1: Comparison: 3 mg Cytisine: Fed vs 3 mg Cytisine: Fasted; Fed/Fasted Ratio; Test type: Superiority; Geometric Least Squares Mean = 79.57, 90% CI 2-sided [66.40 to 95.35]

2. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) Extrapolated to Infinity (AUC0-∞)
Time Frame: Pre-dose (within 60 minutes prior to dosing) up to 48 hours post dose on Days 1-5
Population: PK Set: All randomized participants who received both doses of cytisine and had sufficient, protocol-compliant plasma concentration-time profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
h*ng/mL | 165 (17.5) | 179 (13.7)
Statistical Analysis 1: Comparison: 3 mg Cytisine: Fed vs 3 mg Cytisine: Fasted; Fed/Fasted Ratio; Test type: Superiority; Geometric Least Squares Mean = 92.08, 90% CI 2-sided [88.37 to 95.95]

3. Primary Outcome: Total Cytisine Excreted in Urine Over 48 Hours (Ae0-48h)
Time Frame: Pre-dose (within 60 minutes prior to dosing) up to 48 hours post dose on Days 1-5
Population: Urine Excretion Set: All participants who received both doses of cytisine and had sufficient, protocol-compliant plasma concentration-time profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
mg | 2.40 (21.3) | 2.64 (15.4)
Statistical Analysis 1: Comparison: 3 mg Cytisine: Fed vs 3 mg Cytisine: Fasted; Fed/Fasted Ratio; Test type: Superiority; Geometric Least Squares Mean = 90.89, 90% CI 2-sided [84.99 to 97.20]

4. Primary Outcome: Percent of Total Cytisine Excreted in Urine Over 48 Hours (Ae0-48h%)
Time Frame: Pre-dose (within 60 minutes prior to dosing) up to 48 hours post dose on Days 1-5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of cytisine excreted in urine
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
percent of cytisine excreted in urine | 82.60 (17.627) | 89.22 (13.777)

5. Secondary Outcome: Time to Cmax (Tmax)
Time Frame: Pre-dose (within 60 minutes prior to dosing) up to 48 hours post dose on Days 1-5
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
hours | 1.50 [0.500 to 6.00] | 0.750 [0.333 to 1.50]
Statistical Analysis 1: Comparison: 3 mg Cytisine: Fed vs 3 mg Cytisine: Fasted; Fed/Fasted Ratio; Test type: Superiority; Geometric Least Squares Mean = 1.00, 90% CI 2-sided [0.25 to 1.75]

6. Secondary Outcome: Terminal Elimination Half-Life (T1/2)
Time Frame: Pre-dose (within 60 minutes prior to dosing) up to 48 hours post dose on Days 1-5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
hours | 4.59 (0.566) | 4.73 (0.437)

7. Secondary Outcome: AUC From Time of Dosing to Last Measurable Concentration (AUC0-t)
Time Frame: Pre-dose (within 60 minutes prior to dosing) up to 48 hours post dose on Days 1-5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 12
h*ng/mL | 158 (17.2) | 173 (13.2)
Statistical Analysis 1: Comparison: 3 mg Cytisine: Fed vs 3 mg Cytisine: Fasted; Fed/Fasted Ratio; Test type: Superiority; Geometric Least Squares Mean = 91.40, 90% CI 2-sided [87.55 to 95.41]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Withdrawal of Study Drug
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) is defined as an AE that: results in death; is life-threatening; requires hospitalization or prolongs existing inpatient hospitalization; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; is an important medical event which requires medical intervention to prevent any of the above outcomes. TEAEs are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of investigational product that worsen after the participant receives the first dose of investigational product. Relationship of the TEAE to study drug was evaluated as: definite, probably, possible, unlikely, or not related.
Time Frame: Baseline (Day 0) through Day 5 plus 6-8 days
Population: Safety Set: All randomized participants who received at least 1 dose of cytisine.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 13
Participants
  TEAE | 2 | 0
  Serious TEAE | 0 | 0
  TEAE Leading to withdrawal of study drug | 0 | 0
  Mild TEAE | 2 | 0
  Moderate TEAE | 0 | 0
  Severe TEAE | 0 | 0
  TEAE Relationship: Unlikely | 1 | 0
  TEAE Relationship: Not Related | 1 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Biochemistry, Hematology, Urinalysis, and/or 12-lead Electrocardiogram (ECG) Values
Time Frame: Screening through Day 5
Population: Safety Set: All randomized participants who received at least 1 dose of cytisine.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
Number analyzed (Participants) | 12 | 13
Participants
  Biochemistry | 0 | 0
  Hematology | 0 | 0
  Urinalysis | 0 | 0
  ECG | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) through Day 5 plus 6-8 days
Description: TEAEs are presented
Arm/Group | 3 mg Cytisine: Fed | 3 mg Cytisine: Fasted
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 2/12 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg Cytisine: Fed (N=12) | 3 mg Cytisine: Fasted (N=13)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03509948/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT03509948/SAP_001.pdf